CLINICAL TRIAL: NCT00799695
Title: Diabetic Retina Exam Rate Does Not Increase With Phone Reminders in Non-HMO Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Blue Cross Blue Shield of Michigan Foundation (Other)
Responsible Party: Robert M. Levine, MD, Henry Ford Health System
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: F10030; F10030; 13.13PIRAP
Record Dates: First submitted 2008-11-26; First posted 2008-12-01 (Estimated); Last update posted 2008-12-01 (Estimated); Status verified 2008-11

CONDITIONS: Diabetic Retinopathy
Keywords: diabetic retinopathy; screening; annual
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: phone call contact — A sample of subjects who had not completed their annual diabetic screening exams were contacted by phone and offered appointments for eye exams

SUMMARY:
Diabetic retinopathy is the major cause of blindness in working age Americans, and screening for it is cost-effective. There are a quarter of a million people in Southeast Michigan with diabetes and pre-diabetes.

Only half of patients with diabetes are screened regularly for diabetic retinopathy, and this proportion has been difficult to increase despite various interventions. Previous research focused on HMO patient groups because preventative care was thought to decrease plan costs. In addition, it was administratively feasible to track patient-doctor interactions.

This project builds on published research and institutional experience to determine an effective method for increasing the screening rate, in a mobile, non-HMO population. It uses administrative methods and information technology infrastructures, such as large scale electronic medical records and patient demographic databases, to identify existing patients requiring examinations.

Patients were telephoned by a trained service representative who offered and scheduled firm examination appointment times.

Hypothesis: Annual screening rates for diabetic retinopathy can be substantially improved in non-HMO patient groups by directly contacting patients and scheduling firm appointment times.

ELIGIBILITY:
Inclusion Criteria:

* were Henry Ford Health System patients,
* diabetic
* using the BCBSM payer plan

Exclusion Criteria:

* retina examination in prior year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 561 (Actual)
Dates: Start 2008-01; Primary Completion 2008-05 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
a change in the proportion of diabetic patients who acted as a result of the phone contact, and obtained a retina eye exam. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Levine,, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States